CLINICAL TRIAL: NCT05582629
Title: A Multicenter, Double-blind, Randomized, Placebo-Controlled, Phase III Clinical Study to Evaluate the Efficacy and Safety of JT001 (VV116) in Participants With Mild to Moderate COVID-19
Brief Title: JT001 (VV116) for the Treatment of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JT001-015-III-COVID-19
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Mild to Moderate COVID-19
MeSH Terms: interventions — GS-621763

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): JT001 (VV116) Day 1: 0.6g, Q12H X 2 times Day 2-5: 0.3g, Q12H X 8 times Oral tablet
  Interventions: Drug: JT001
- Arm 2 (Placebo Comparator): Placebo Day 1: 6 tablets, Q12H X 2 times Day 2-5: 3 tablets, Q12H X 8 times Oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JT001 — JT001 administered orally in tablet form every 12 hours for 5 days
  Other Names: VV116
  Arms: Arm 1
Drug: Placebo — Placebo matching JT001 administered orally in tablet form every 12 hours for 5 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JT001 (VV116) in participants with mild to moderate COVID-19.

DETAILED DESCRIPTION:
Screening Interested participants will sign the appropriate informed consent form (ICF) prior to completion of any study procedures.

The investigator will review symptoms and other non-invasive inclusion and exclusion criteria prior to any invasive procedures. If the participant is eligible after this review, then the site will perform the invasive procedures to confirm eligibility.

Treatment and Assessment

This is the general sequence of events during the 28-day treatment and assessment period:

Complete baseline procedures and samples collection； Participants are randomized to experimental arm or placebo arm； Participants receive study intervention (Q12H X 5 days)； Complete all safety monitoring； Complete all efficacy data collection； Blood samples collection

ELIGIBILITY:
Inclusion Criteria:

1. Participants of 18 years of age or older, at the time of signing of informed consent.
2. Have a positive SARS-CoV-2 test result, and sample collection for the first positive SARS-CoV-2 viral infection determination ≤5 days prior to the first dose.

   Note: PCR is the preferred method; however, with evolving approaches to laboratory confirmation of SARS-CoV-2 infection, other molecular or antigen tests that detect viral RNA or protein are allowed if authorized for use in the country. Serological tests that detect host antibodies generated in response to recent or prior infection are not allowed.
3. Initial onset of symptoms of COVID-19 ≤3 days prior to the first dose.
4. Have any of the following targeted COVID-19-related symptoms with COVID-19 Related Symptoms score ≥2 within 24 hours before the first dose:

   fever

   cough

   sore throat

   stuffy or running nose,

   headache

   muscle or body aches

   shortness of breath or difficulty breathing

   nausea

   chills or shivering

   vomiting

   diarrhea
5. Agree to adhere to contraception restrictions.Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
6. Understand and agree to comply with planned study procedures.
7. Can give written informed consent approved by the Ethical Review Board governing the site and comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Severe or critical COVID-19.
2. SpO2≤93% on room air at sea level or PaO2/FiO2≤ 300 (with oxygen inhalation), or respiratory rate ≥30 per minute, or heart rate ≥125 per minute.
3. Require mechanical ventilation or anticipated impending need for mechanical ventilation.
4. Are suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention.
5. Current eye disease (such as inflammation, vessel deformity, retinal hemorrhage or decollement, optic nerve lesion, or fundus lesion).
6. ALT or AST>2 ULN at screening.
7. Allergies to any of the components used in the formulation of the interventions.
8. Any medical condition, which in the opinion of the Investigator, will compromise the safety of the participant.
9. Received a SARS-CoV-2 monoclonal antibody treatment or prevention, or antiviral treatment (including the investigational treatment) within 30 days prior to screening.
10. Received convalescent COVID-19 plasma treatment within 30 days prior to screening.
11. Participated in a clinical study involving an investigational intervention within the last 30 days. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
12. Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
13. Female who are pregnant or breast-feeding or plan to be pregnant within this study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Characterize the effect of JT001 (VV116) compared to placebo on clinical recovery | Up to 28 days
  Time to sustained clinical symptoms resolution

SECONDARY OUTCOMES:
Clinical alleviation | Up to 28 days
  Time to sustained clinical symptoms alleviation
Disease progression | Up to 28 days
  Percentage of participants who experience the following events of disease progression through Day 28 COVID-19-related hospitalization in non-hospitalized participants Progression to severe COVID-19 Progression to critical COVID-19 Death from any cause
SARS-CoV-2 nucleic acid and viral load | Up to 28 days
  Percentage of participants who achieve SARS-CoV-2 negative through Days 5 and 7 Change of SARS-CoV-2 Ct Value from baseline to Days 5 and 7 Change of SARS-CoV-2 viral load from baseline to Days 5 and 7 SARS-CoV-2 viral load area under the response time curve (AUC) assessed through Day 7
Safety | Up to 28 days
  Safety assessments such as AEs and SAEs through Day 28

OTHER OUTCOMES:
SARS-CoV-2 viral genetic variation | Day 1
  To assess SARS-CoV-2 viral genetic variation
SARS-CoV-2 negative | Up to 28 days
  Time to SARS-CoV-2 negative

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Fuzhou Pulmonary Hospital Of Fujian, Fuzhou, Fujian
  - The third people's hospital of Shenzhen, Shenzhen, Guangdong
  - Wuhan Infections Diseases Hospital, Wuhan, Hubei
  - The Fourth Hospital in Inner Mongolia, Hohhot, Inner Mongolia
  - The Sixth People's Hospital of ShenYang, Shenyang, Liaoning
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol
Time Frame: With publication :
  Access to all individual participant data collected during the trial, will be provided after anonymization with publication.No expiration date of data requests is currently set once data are made available. Access is provided after a proposal has been approved by an independent review committee identified for this purpose and after receipt of a signed data sharing agreement. Data and documents will be provided in a secure data sharing environment.
Access Criteria: Upon request to the corresponding authors (ljli@zju.edu.cn). Qualified science and medical researchers upon formal request and submission of research proposal detailing planned analyses.
  De-identified individual participant data and relevant clinical trial documents will be shared for the purpose of conducting legitimate research as specified in an approved formal research proposal.

REFERENCES:
- [Derived] Fan X, Dai X, Ling Y, Wu L, Tang L, Peng C, Huang C, Liu H, Lu H, Shen X, Zhang W, Wang F, Li G, Li M, Huang Y, Zhang H, Li M, Ren F, Li Y, Liu C, Zhou Z, Sun W, Yi Y, Zhou D, Gao H, Pan Q, Liu H, Zhao J, Ding Z, Ma Y, Li W, Wang Q, Wang X, Bai Y, Jiang X, Ma J, Xie B, Zhang K, Li L. Oral VV116 versus placebo in patients with mild-to-moderate COVID-19 in China: a multicentre, double-blind, phase 3, randomised controlled study. Lancet Infect Dis. 2024 Feb;24(2):129-139. doi: 10.1016/S1473-3099(23)00577-7. Epub 2023 Nov 22. PMID 38006892